CLINICAL TRIAL: NCT01576289
Title: Clinical Evaluation and Histological Analysis of Biopsies From the Upper Gastrointestinal Tract of Patients With and Without Symptoms of Reflux Disease (histoGERD Trial)
Brief Title: Analysis of Biopsies From the Upper Gastrointestinal Tract
Acronym: histoGERD
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Cord Langner, MD, MD, Senior Scientist, Medical University of Graz
Other Study IDs: Reflux_Multicenter_1
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux Disease; Gastritis
Keywords: Esophagus; Gastroesophageal reflux; Reflux esophagitis; Barrett's esophagus; Stomach; Intestinal metaplasia stomach; Helicobacter pylori infection; Proton pump inhibitor; Duodenum; Duodenal bulb; Celiac disease diagnosis
MeSH Terms: conditions — Gastroesophageal Reflux; Gastritis; Esophagitis, Peptic; Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy specimens (formalin fixed and paraffin embedded) which are routinely obtained during the endoscopic procedure are retained according to legal requirements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing uppper endoscopy: Consecutive patients with and without symptoms of reflux disease who routinely undergo upper endoscopy from November 2011 through May 2012.
  Interventions: Other: Histological analysis

INTERVENTIONS:
Other: Histological analysis — Systematic histological analysis of biopsy specimens obtained during routine endoscopic examination

SUMMARY:
Multicenter study to correlate histological findings in the upper gastrointestinal tract with endoscopic and clinical data.

DETAILED DESCRIPTION:
Prospective multicenter study involving six clinical institutions (see collaborators) with recruitment of consecutive patients who undergo routine upper endoscopy for several (non-selected) reasons. The patients will have to fill out a questionnaire about their history of reflux symptoms, including questions regarding smoking and drinking habits. The treating physician will have to complete a clinical protocol which includes a questionnaire regarding the patient's drug history.

The endoscopic examination is done in a routine, yet standardized fashion. In particular, biopsy material will be taken from the stomach, the gastroesophageal junction and from the duodenum. The samples will be routinely sent to the participating institutes of pathology (see collaborators) and will be assessed by independent histopathologists with special expertise in gastrointestinal pathology.

Endoscopic findings are documented in a standardized clinical protocol. Likewise, the histopathological assessment of the samples is done following a standardized protocol following the WHO classification and the updated Sydney classification, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* Patients with abnormal anatomy at the gastroesophageal junction (e.g. post surgery)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who routinely undergo upper endoscopy (for different, not selected reasons)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cord Langner, MD, Principal Investigator — Medical University of Graz, Institute of Pathology, A 8036 Graz, Austria
Locations (1):
- Medical University, Graz, Austria